CLINICAL TRIAL: NCT00251862
Title: Shared Decision-Making for Colorectal Cancer Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 5R01HS013912-05 (AHRQ)
Record Dates: First submitted 2005-11-09; First posted 2005-11-11 (Estimated); Results first posted 2013-12-02 (Estimated); Last update posted 2013-12-27 (Estimated); Status verified 2013-09

CONDITIONS: Colorectal Cancer
Keywords: Colorectal cancer screening; Shared decision-making; Decision aid
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Decision Support Techniques

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- Decision aid plus YourDiseaseRisk (Experimental): Patients viewed the decision aid and completed the Your Disease Risk risk assessment tool prior to visit with their primary care provider.
  Interventions: Behavioral: Web-based decision aid plus personalized risk assessment
- Decision aid alone (Experimental): Patient's viewed decision aid only prior to a visit with their primary care provider.
  Interventions: Behavioral: Web-based decision aid alone
- III (Sham Comparator): Standard care
  Interventions: Behavioral: Generic website

INTERVENTIONS:
Behavioral: Web-based decision aid plus personalized risk assessment — Patients review a computer-based decision aid that discuss the pros and cons of of 5 recommended CRC screening options and provides personalized 10-year estimates of CRC risk prior to meeting with their provider to discuss CRC screening.
  Other Names: Decision aid, personalized risk assessment tool
  Arms: Decision aid plus YourDiseaseRisk
Behavioral: Web-based decision aid alone — Patients review a computer-based decision aid that discuss the pros and cons of the 5 recommended CRC screening options prior to meeting with their provider to discuss CRC screening.
  Other Names: Decision aid
  Arms: Decision aid alone
Behavioral: Generic website — Patients review a generic website that discuss ways to reduce overall cancer risk.
  Other Names: Control condtion
  Arms: III

SUMMARY:
The overall objective of this study is to conduct a three-arm randomized controlled trial to evaluate the impact of an interactive, web-based decision aid on shared decision-making and patient adherence to colorectal cancer (CRC) screening recommendations.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the second leading cause of cancer-related death and third most commonly diagnosed cancer among men and women in the United States. Screening has been shown to be a cost-effective strategy for reducing both CRC mortality through early detection and incidence through the detection and removal of precancerous adenomatous polyps (adenomas). Despite a compelling rationale and widespread endorsement by authoritative groups, screening rates remain far below those necessary to achieve significant reductions in CRC mortality or incidence. Poor patient acceptance and non-adherence to screening recommendations are partly responsible for low screening rates. Shared decision-making has been advocated as a potentially effective yet unproven strategy for addressing this problem. Implicit in this approach is the need for an unbiased decision aid that not only educates patients about the pros and cons of the different strategies so as to enable them to identify a preferred strategy but also empowers patients to take a proactive role in the decision-making process, thereby increasing satisfaction and promoting adherence. From a logistical standpoint, the decision aid must also be easy to implement in the ambulatory setting so as to maximize use but minimize demands on physician time and office resources. To address this need, we have developed an interactive, web-based decision aid and implementation strategy for use in routine clinical practice.

Comparison(s): Average risk subjects assigned to one of two intervention arms (decision aid alone versus decision aid plus personalized risk assessment with feedback) compared to a control arm(generic website that discusses lifestyle changes that can reduce overall cancer risk).

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic average-risk subjects
* Under the direct care of one of participating site's staff (attending) physicians or physician extenders;
* No prior screening other than fecal occult blood testing (FOBT);
* No major co-morbidities that preclude CRC screening by any method

Exclusion Criteria:

* Prior CRC screening by any method other than FOBT occult blood testing
* High-risk condition (personal history of colorectal cancer or polyps, family history of colorectal cancer or polyps involving one or more first degree relatives, chronic inflammatory bowel disease)
* Lack of fluency in written and spoken English (since decision aid and personalized risk assessment tool will be in English only due to funding issues);
* Comorbidities that preclude CRC screening by any method

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 825 (Actual)
Dates: Start 2005-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul C. Schroy III, MD, MPH, Principal Investigator — Boston Medical Center
Locations (2):
- United States (2):
  - Boston Medical Center, Boston, Massachusetts
  - South Boston Community Health Center, Boston, Massachusetts

REFERENCES:
- [Background] Schroy PC 3rd, Glick JT, Robinson PA, Lydotes MA, Evans SR, Emmons KM. Has the surge in media attention increased public awareness about colorectal cancer and screening? J Community Health. 2008 Feb;33(1):1-9. doi: 10.1007/s10900-007-9065-5. PMID 18080203
- [Background] Schroy PC 3rd, Glick JT, Robinson P, Lydotes MA, Heeren TC, Prout M, Davidson P, Wong JB. A cost-effectiveness analysis of subject recruitment strategies in the HIPAA era: results from a colorectal cancer screening adherence trial. Clin Trials. 2009 Dec;6(6):597-609. doi: 10.1177/1740774509346703. Epub 2009 Nov 23. PMID 19933718
- [Background] Schroy PC 3rd, Mylvaganam S, Davidson P. Provider perspectives on the utility of a colorectal cancer screening decision aid for facilitating shared decision making. Health Expect. 2014 Feb;17(1):27-35. doi: 10.1111/j.1369-7625.2011.00730.x. Epub 2011 Sep 8. PMID 21902773
- [Result] Schroy PC 3rd, Emmons K, Peters E, Glick JT, Robinson PA, Lydotes MA, Mylvanaman S, Evans S, Chaisson C, Pignone M, Prout M, Davidson P, Heeren TC. The impact of a novel computer-based decision aid on shared decision making for colorectal cancer screening: a randomized trial. Med Decis Making. 2011 Jan-Feb;31(1):93-107. doi: 10.1177/0272989X10369007. Epub 2010 May 18. PMID 20484090
- [Result] Schroy PC 3rd, Emmons KM, Peters E, Glick JT, Robinson PA, Lydotes MA, Mylvaganam SR, Coe AM, Chen CA, Chaisson CE, Pignone MP, Prout MN, Davidson PK, Heeren TC. Aid-assisted decision making and colorectal cancer screening: a randomized controlled trial. Am J Prev Med. 2012 Dec;43(6):573-83. doi: 10.1016/j.amepre.2012.08.018. PMID 23159252

RESULTS

PARTICIPANT FLOW:
Groups:
- DA + YDR: Decision aid (DA) plus Your Disease Risk (YDR) personalized risk feedback
- DA Alone: Decision aid alone
- Control: Standard Care
Period: Overall Study
Arm/Group | DA + YDR | DA Alone | Control
Started | 280 | 269 | 276
Completed | 280 | 269 | 276
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DA + YDR | DA Alone | Control | Total
Number analyzed (Participants) | 280 | 269 | 276 | 825
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 232 | 234 | 230 | 696
  >=65 years | 48 | 35 | 46 | 129
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 163 | 164 | 159 | 486
  Male | 117 | 105 | 117 | 339
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 10 | 15 | 43
  Not Hispanic or Latino | 262 | 259 | 261 | 782
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 7 | 2 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 172 | 160 | 180 | 512
  White | 99 | 96 | 88 | 283
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 6 | 6 | 6 | 18
Region of Enrollment [Number; unit: participants]
  United States | 280 | 269 | 276 | 825

OUTCOME MEASURES:

1. Primary Outcome: Patient Adherence (Test Completion)
Description: Completion of a screening test within 12 months of the study visit.
Time Frame: 12 months post-intervention
Population: Intention to treat
Measure: Number; unit: participants
Arm/Group | DA + YDR | DA Alone | Control
Number analyzed (Participants) | 280 | 269 | 276
participants | 104 | 116 | 96
Statistical Analysis 1: Comparison: DA + YDR vs Control; Sample size and power considerations focused on a two-group comparison of the DA alone versus control study arms for the primary outcome of colorectal cancer (CRC) screening test completion at 12 months. Based on crude estimates of baseline test completion rates, we calculated that a target sample of 275 subjects per arm provided greater than 80% power of detecting a 54% vs. 40% difference at the P<0.05 level; Test type: Superiority or Other; p = 0.046, Chi-squared; Absolute Difference = 8.3, 95% CI 2-sided [-2.2 to 14.2]
Statistical Analysis 2: Comparison: DA + YDR vs DA Alone; Test type: Superiority or Other; p = 0.153, Chi-squared; Absolute Difference = 6.0, 95% CI 2-sided [0.2 to 16.5]

2. Secondary Outcome: Patient Knowledge
Description: Knowledge was assessed at baseline (pretest) and at the time of the exit survey (posttest) based on responses to a 12-item questionnaire (True/False/Don't know) that inquired about CRC risk factors, the rationale and goals of screening, and age at which screening should begin. Cumulative knowledge scores (range, 0-12) were derived by summing correct responses to the 12 individual knowledge questions.
Time Frame: Immediate post-intervention study visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DA + YDR | DA Alone | Control
Number analyzed (Participants) | 280 | 269 | 276
units on a scale | 10.7 (1.9) | 10.9 (1.6) | 8.6 (2.6)
Statistical Analysis 1: Comparison: DA + YDR vs DA Alone vs Control; The three study groups were compared on cumulative pre-test and post-test knowledge through separate one-factor analysis of covariance (ANCOVA); followed pairwise comparisons using Bonferroni's adjusted multiple comparison procedure; Test type: Superiority or Other; p < 0.001, ANCOVA — Pairwise comparisons: DA+YDR vs. Control, P<0.001; DA alone vs. Control, P<0.001

3. Secondary Outcome: Patient Satisfaction With Decision Making Process
Description: Patient satisfaction with the decision-making process (SDMP) was assessed using the validated 12-item Satisfaction with the Decision-Making Process scale. Five ordered response categories were used for each item. Each response was assigned a point score ranging from 1 for "strongly disagree" (or "poor") to 5 for "strongly agree" (or "excellent"). A cumulative score was calculated based on the summed response scores for each item (maximum score = 60). Mean item substitution was used to impute missing data.
Time Frame: Immediate post-intervention primary care provider (PCP) visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DA + YDR | DA Alone | Control
Number analyzed (Participants) | 280 | 269 | 276
units on a scale | 49.0 (6.2) | 49.7 (6.4) | 45.5 (7.8)
Statistical Analysis 1: Comparison: DA + YDR vs DA Alone vs Control; The three study groups were compared through separate one-factor analysis of covariance (ANCOVA); followed pairwise comparisons using Bonferroni's adjusted multiple comparison procedure; Test type: Superiority or Other; p < 0.001, ANCOVA

4. Secondary Outcome: Screening Intentions
Description: Screening intentions were also assessed as part of the posttest. Subjects were asked how sure they were that they would schedule an appointment to get screened for colorectal cancer and how sure they were that they would complete the screening test they scheduled. An ordered 5-point response frame was used ranging from 1 for "not at all sure" to 5 for "completely sure".
Time Frame: Immediate post-intervention study visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DA + YDR | DA Alone | Control
Number analyzed (Participants) | 280 | 269 | 276
units on a scale | 4.4 (1.0) | 4.4 (1.0) | 4.0 (1.3)
Statistical Analysis 1: Comparison: DA + YDR vs DA Alone vs Control; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA

ADVERSE EVENTS:
Arm/Group | DA + YDR | DA Alone | Control
Serious Adverse Events (participants affected / at risk) | 0/280 | 0/269 | 0/276
Other Adverse Events (participants affected / at risk) | 0/280 | 0/269 | 0/276

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes